CLINICAL TRIAL: NCT02601807
Title: A Randomised Controlled Trial to Assess the Benefits of ActiPatch-Pulsed Shortwave Therapy for Chronic Lower Back Pain
Brief Title: ActiPatch Therapy for Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15/LO/0926
Record Dates: First submitted 2015-10-21; First posted 2015-11-10 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Back Ache
Keywords: Back; Pain; PSWT; ActiPatch; Pulsed shortwave therapy
MeSH Terms: conditions — Back Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Active Comparator): Subjects given active ActiPatch device before or after crossover (randomised)
  Interventions: Device: ActiPatch (active)
- Placebo (Placebo Comparator): Subjects given placebo ActiPatch device before or after crossover (randomised)
  Interventions: Device: ActiPatch (placebo)

INTERVENTIONS:
Device: ActiPatch (active) — Active version of the ActiPatch pulsed shortwave therapy device. Emits shortwave radiofrequency pulsed energy.
  Other Names: Pulsed shortwave therapy (placebo)
  Arms: Active
Device: ActiPatch (placebo) — Placebo version of the ActiPatch pulsed shortwave therapy device. Emits no radiofrequency energy but otherwise appears identical to the active device.
  Other Names: Pulsed shortwave therapy (active)
  Arms: Placebo

SUMMARY:
The ActiPatch is a cutaneous device which is CE marked approved for relief of pain. It is taped over the affected area and stimulation at a high frequency is reported to alleviate pain with no sensation. However there is no class 1 evidence for this on back pain. By randomising patients between application of an active device or a dummy device and assessment of disability and pain scores at two weeks, the efficacy or otherwise can be established. Low back pain is a major health problem and if effective this has major economic implications as the device is cheap and safe.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.
* Male or female ages 18-90 years old with stable chronic low back pain
* ≥3 months duration of chronic low back pain
* a current VAS pain rating ≥5/10
* no radiating pain below the knee
* ≥75% back or buttock pain rather than lower extremity pain
* Able to complete and tolerate treatment for the study period.

Exclusion Criteria:

* Female participant who is pregnant
* Significant renal or hepatic impairment.
* Prior home use of pulsed shortwave therapy
* Prior history of spinal fusion or failed spinal surgery syndrome.
* Laminectomy, laminotomy or discectomy within 12 months of enrollment.
* Diagnostic or interventional injections or any low back surgeries not mentioned above, including radiofrequency neuroablation within 6 months of enrollment.
* Any addition of strong opiates, pregabalin and gabapentin to the treatment regime during the course of the trial
* Current implanted cardiac demand pacemakers, defibrillators, cardiac pumps, spinal stimulators or other implanted electronic devices.
* Patients using personal home based electrical stimulation devices
* Patients with other concomitant illnesses (e.g., malignancy, osteoporosis) which, in the opinion of the investigator, would preclude successful patient participation will also be excluded
* Active psychiatric disorders (as evidenced by use of antipsychotic or medication).
* Patients diagnosed with history of significant mood disorder will be excluded (depression or anxiety with adequate control would be acceptable).
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Participant with life expectancy of less than 6 months, or inappropriate for placebo medication.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks.
* Participants who are not able to understand verbal or written English, and for whom adequate translation/interpretation cannot be readily obtained.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Pain-related disability, indexed by the Oswestry Disability Index (ODI) | Change from baseline ODI score at 2 weeks

SECONDARY OUTCOMES:
Subjective pain, indexed by Visual analogue pain scale | Change from baseline visual analogue score over the course of 2 weeks, recorded daily during the 2 week period by participant as part of a pain diary
Medication intake | Change from baseline medication intake rate over the course of 2 weeks, recorded daily during the 2 week period by participant as part of a pain diary
Pain related disability, indexed by the Roland Morris Instrument | Change from baseline Roland Morris Instrument scores at 2 weeks
Quality of life, indexed by the EQ-5D-5L questionnaire | Change from baseline EQ-5D-5L scores at 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom